CLINICAL TRIAL: NCT02080819
Title: Striatal Effective Connectivity to Predict Treatment Response in Cocaine Misuse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM20000079; 1R01DA034131 (NIH); PT109865 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Results first posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-03

CONDITIONS: Cocaine Dependence
Keywords: drug abuse; cocaine; impulsivity; dopamine
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders; Impulsive Behavior | interventions — Levodopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy Control (No Intervention): Non drug using healthy controls
- Placebo (Placebo Comparator): Placebo BID for 7 weeks
  Interventions: Drug: levodopa/carbidopa 400/100 BID
- Medication (Experimental): Levodopa/carbidopa 400/100 BID for 7 weeks
  Interventions: Drug: levodopa/carbidopa 400/100 BID

INTERVENTIONS:
Drug: levodopa/carbidopa 400/100 BID — Levodopa dose escalation (1 week): Days 1-2, one 50/12.5 mg tablet BID; Days 3-4, one 100/25 mg tablet BID; Days 5-6, one 200/50 mg tablet BID; Day 7, one 400/100 mg tablet BID.
  Maintenance phase (7 weeks): One 400/100 mg Levodopa/Carbidopa tablet BID or placebo in conjunction with once weekly individual cognitive behavioral therapy plus contingency management for attendance.
  Other Names: Sinemet; Parcopa
  Arms: Medication; Placebo

SUMMARY:
This project proposes to investigate the role of brain connectivity in the mechanism of treatment response to dopaminergic medications in cocaine dependence.

DETAILED DESCRIPTION:
This project will use stochastic DCM, which is a recent DCM extension that takes into account hidden fluctuations in neuronal and vascular responses, and thus is especially suited for investigating effects of disease or drugs. In addition, this project will use nonlinear DCM, a DCM extension that can measure gating effects by striatum on cortico-cortical pathways. The overall aims of this project are: (1) To conduct functional magnetic resonance imaging-based DCM studies of working memory and impulsivity in order to determine the effective (directional) connectivity between PFC and striatum in treatment-seeking Cocaine Dependent (CD) subjects compared to non-drug using controls. We hypothesize that DLPFC causally affects ventral striatum in CDs, and that the strength of this connection is lower in CDs compared to controls. (2) To determine whether the pretreatment gating effect by the dorsal striatum, as a reflection of pretreatment hypodopaminergic state associated with chronic compulsive drug use, predicts the treatment response to dopaminergic pharmacotherapy in CDs. We hypothesize that lower pretreatment gating by the dorsal striatum on prefrontal-parietal effective connectivity predicts greater 8-week improvement from treatment of CDs with DA enhancing medications (combined with cognitive behavioral therapy [CBT]), but not from treatment with placebo (combined with CBT).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Age 18 to 50
* Meet current DSM-IV criteria for cocaine dependence who are seeking treatment.

Exclusion Criteria:

1. Current DSM-IV diagnosis of any psychoactive substance dependence other than cocaine, marijuana, nicotine, or alcohol
2. Have a DSM-IV axis I psychiatric disorder or neurological disease or disorder requiring ongoing treatment and/or making study participation unsafe
3. Significant current suicidal or homicidal ideation
4. Medical conditions contraindicating levodopa/carbidopa or pharmacotherapy (e.g., evidence of any movement disorder, clinically significant pulmonary disease, cardiovascular disease, liver or kidney disease, seizure disorder)
5. Taking CNS active concomitant medications
6. Taking medications known to have significant drug interactions with the study medication (e.g., CYP P-450-2D6 inhibitors, such as tamoxifen, iron salts, pyridoxine, monoamine oxidase inhibitors, phenothiazines, selegiline, anesthetics)
7. Having conditions of probation or parole requiring reports of drug use to officers of the court
8. Impending incarceration
9. Pregnant or breast feeding for female patients
10. Inability to read, write, or speak English
11. Having plans to leave the immediate geographical area within 3 months
12. Unwillingness or not competent to sign a written informed consent form
13. Individuals who have pacemakers, metal or electromechanical implants or metallic foreign bodies
14. Patients who are known to be HIV positive will not be included due to possible CNS effects of HIV.
15. Alcohol withdrawal symptoms or history of significant previous alcohol withdrawal symptoms

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2014-02; Primary Completion 2017-01-21 (Actual); Study Completion 2017-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liangsuo Ma, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo BID for 7 weeks
  levodopa/carbidopa 400/100 BID: Levodopa dose escalation (1 week): Days 1-2, one 50/12.5 mg tablet BID; Days 3-4, one 100/25 mg tablet BID; Days 5-6, one 200/50 mg tablet BID; Day 7, one 400/100 mg tablet BID.
  Maintenance phase (7 weeks): One 400/100 mg Levodopa/Carbidopa tablet BID or placebo in conjunction with once weekly individual cognitive behavioral therapy plus contingency management for attendance.
- Medication: Levodopa/carbidopa 400/100 BID for 7 weeks
  levodopa/carbidopa 400/100 BID: Levodopa dose escalation (1 week): Days 1-2, one 50/12.5 mg tablet BID; Days 3-4, one 100/25 mg tablet BID; Days 5-6, one 200/50 mg tablet BID; Day 7, one 400/100 mg tablet BID.
  Maintenance phase (7 weeks): One 400/100 mg Levodopa/Carbidopa tablet BID or placebo in conjunction with once weekly individual cognitive behavioral therapy plus contingency management for attendance.
Period: Overall Study
Arm/Group | Healthy Control | Placebo | Medication
Started | 63 | 35 | 33
Completed | 38 | 9 | 11
Not Completed | 25 | 26 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Control | Placebo | Medication | Total
Number analyzed (Participants) | 38 | 9 | 11 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 38 | 9 | 11 | 58
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (12) | 33 (7) | 35 (8) | 33 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 4 | 1 | 24
  Male | 19 | 5 | 10 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 0 | 3
  Black or African American | 21 | 9 | 10 | 40
  White | 9 | 0 | 1 | 10
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 38 | 9 | 11 | 30

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Treatment Outcome
Description: Treatment effectiveness score based on number of positive urine drug screens
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: positive drug screens
Arm/Group | Healthy Control | Placebo | Medication
Number analyzed (Participants) | 38 | 9 | 11
positive drug screens | 0 (0) | 14 (15) | 13 (9)

ADVERSE EVENTS:
Arm/Group | Healthy Control | Placebo | Medication
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/38 | 0/9 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-10-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT02080819/Prot_000.pdf
  • Statistical Analysis Plan (2013-10-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT02080819/SAP_001.pdf